CLINICAL TRIAL: NCT04146025
Title: Leveraging Urban Nature, Behavioral Economics, and Mobile Platforms to Prevent Postpartum Depression
Brief Title: Nurtured in Nature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 833693
Record Dates: First submitted 2019-10-02; First posted 2019-10-31 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Postpartum Depression; Pregnancy Related; Environmental Exposure
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature Coach Intervention (Experimental): The Nature Coach Intervention consists of 3 components - home visit, text message follow up, and goal feedback.
  Interventions: Behavioral: Nature Coach Intervention
- Control Group (No Intervention): Education only

INTERVENTIONS:
Behavioral: Nature Coach Intervention — 1. Home visit. During the 1-hour home visit, the coach will (a) provide education about the health benefits of nature, (b) identify nearby nature targets for the participant to visit, (c) complete a pre-commitment contract based on individualized weekly nature goals, and (d) brainstorm barriers and solutions to reaching the goals.
  2. Personalized weekly text messages. Texts will serve as reminders of goals set with the Nature Coach, as well as encouragement to meet the goals. The context of text messages with change slightly based on individual participants, the goals they set, and the barriers they identify.
  3. Goal feedback- At the end of each week, participants will receive a progression badge via text message that shows the amount of days and time they spent in nature, and how this matched up to the goal set with the Nature Coach.
  Arms: Nature Coach Intervention

SUMMARY:
The investigators pilot test a Nature Coach Intervention in a population of postpartum women, to increase the amount of time people spend outside in local nature, with the goal of preventing postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression (PPD), characterized by feelings of sadness, irritability, and fatigue following the birth of a child, occurs in 10-15% of women. PPD peaks within the first 2-3 months following delivery, but can occur anytime in the first year, representing one of the most common complications of childbearing. The consequences go beyond impaired functioning for the woman, and include harmful effects on the cognitive and emotional development of the woman's infant. Despite this, many women are undiagnosed and do not get adequate treatment.

Living near and spending time in green space is associated with a host of mental health benefits, including reduced depression and improved well-being. Research has shown that women who live near more green space have improved birth outcomes such as higher birthweight infants.

Despite the growing body of evidence linking nature with improved mental health, spending time in green space is not a standard health promoting tool to address mental illness. Behavioral economics concepts have been used successfully in promoting other preventative health behaviors such as physical activity and healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Delivery of a living child
* Ambulatory
* Live in West or Southwest Philadelphia
* Have a smart phone
* Able to understand and respond to an oral interview in English

Exclusion Criteria:

* Baby in Neonatal Intensive Care Unit
* Mother has not been in Intensive Care Unit pre/post-delivery
* Gestational age less than 37 weeks
* Department of Human Services involvement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postpartum women living in West and South West Philadelphia
Enrollment: 36 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Green space use | 3 months
  This will be measured using Global Positioning System (GPS) data to see the amount of time spent in green space.

SECONDARY OUTCOMES:
Prevention of postpartum depression | 3 months
  This will be measured using the Edinburgh Postnatal Depression Scale. The Edinburgh Postnatal Depression Scale is a 10-statement scale that was developed to identify women who may have postpartum depression. Each answer is given a score of 0 to 3.The maximum score is 30
  Questions 1, 2, & 4 are scored 0, 1, 2 or 3 with the first choice option scored as a 0 and the last choice option scored as 3. Questions 3, 5-10 are reverse scored, with the first choice option scored as a 3 and the last choice option scored as a 0. A score of 10 or more suggests that minor or major depression may be present.
Improvement in general well-being | 3 months
  This will be measured using the World Health Organization-5 (WHO-5) Well-being Index. The WHO-5 Well-Being Index is a questionnaire that measures current mental well-being,with the time frame being the previous two weeks.This is five items rated on 6-point Likert scale (All of the time, Most of the time, More than half the time, Less than half the time, Some of the time, At no time). The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia South, MD MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No